CLINICAL TRIAL: NCT05536102
Title: A Single-arm, Open-label, Multicenter Phase 2 Study to Evaluate XELOX + Tislelizumab in Combination With Doxorubicin Hydrochloride Liposome Injection （XELOX+PD-1+PLD）as Neoadjuvant Therapy for Resectable Gastric Cancer
Brief Title: The Effectiveness and Safety of XELOX and Tislelizumab + PLD for Resectable Gastric Cancer (LidingStudy)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qi Li, Chief Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-GC-04
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Gastric Cancer
Keywords: PLD; resectable; XELOX; PD-1
MeSH Terms: conditions — Stomach Neoplasms | interventions — 1-dodecylpyridoxal; liposomal doxorubicin; Oxaliplatin; Capecitabine; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment group (Experimental): Pegylated Liposomal Doxorubicin + Oxaliplatin + Capecitabine + Tislelizumab; reapt every 21 days.
  Interventions: Drug: PLD; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Tislelizumab

INTERVENTIONS:
Drug: PLD — 20mg/m2, day 1, q3w
  Other Names: Pegylated Liposomal Doxorubicin
Drug: Oxaliplatin — 130 mg/m2, day 1, q3w
  Other Names: Eloxatin
Drug: Capecitabine — 1000 mg/m2, days 1-14, q3w
  Other Names: Xeloda
Drug: Tislelizumab — 200 mg, day 1, q3w
  Other Names: BGB-A317

SUMMARY:
This is a signle-arm, multi-center, open-lable, phase II study. The objective is to evaluate the effectiveness and safety of tislelizumab + oxaliplatin + capecitabine + PLD in the neoadjuvant treatment of resectable gastric adenocarcinoma.

DETAILED DESCRIPTION:
This single-arm, multicenter, open-label study plan to enroll patients with resectable stage III gastric adenocarcinoma to recieve tislelizumab + oxaliplatin + capecitabine + PLD regimen for 2 or 4 cycles, radical resection will be performed after neoadjuvant therapy. Radiological evaluation will be performed every 2 cycles to evaluate the resectability of tumor. Survival follow-up will be performed after surgery, until patient's withdrawal of informed consent, loss to follow-up or death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18~75 years old.
2. Karnofsky Performance Status Score ≥70.
3. Histological or cytological diagnosed as gastric adenocarcinoma, HER2-, PD-1/L1+.
4. Clinical stage stage III (8th edition of the AJCC Cancer Staging Manual).
5. Physical condition and organ function allow for larger abdominal surgery.
6. Subject baseline blood routine and biochemical indicators meet the following standards: hemoglobin ≥90g/L; absolute neutrophil count (ANC) ≥1.5×10^9g/L; platelets counts (PLT) ≥100×10^9/L; alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal (ULN); serum total bilirubin <1.5 ULN; serum creatinine <1 ULN; serum albumin ≥30g/L.
7. Heart function:

   1. Left ventricular ejection fraction (LVEF) ≥50%;
   2. 12-ECG indicates no myocardial ischemia;
   3. No history of arrhythmia requiring drug intervention before enrollment;
8. No serious concomitant diseases that make the survival time < 5 years.
9. Agree and be able to comply with the protocol during the study period.
10. Provide written informed consent before entering the study.

Exclusion Criteria:

1. Received chemotherapy, radiotherapy or immunotherapy for this gastric cancer.
2. Pregnant or breastfeeding women.
3. Women of childbearing age who had a positive pregnancy test at baseline or who did not have a pregnancy test. Menopausal women must have menopause for at least 12 months before they can become pregnant.
4. Men and women who are sexually active (possible to have children) are unwilling to use contraception during the study period.
5. Patients with mass ascites and positive abdominal free cancer cells.
6. With a history of other malignancies in the last 5 years, except for cured non-melanoma skin cancer and cervical carcinoma in situ.
7. With a history of epilepsy, central nervous system disease, or mental disorder may be judged by the investigator that their clinical severity may hinder the signing of informed consent or affect the patient's oral medication compliance.
8. Clinically severe (i.e. active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) grade II or more severe congestive heart failure, or severe arrhythmia requiring medical intervention, or the last 12 There was a history of myocardial infarction within months.
9. Patients deficiency of dihydropyrimidine dehydrogenase (DPD).
10. Peripheral nerve disease ≥ NCI CTC AE grade 2. However, the patients only with deep tendon reflex (DTR) disappears do not need to be excluded.
11. Organ transplantation requires immunosuppressive therapy.
12. Severe uncontrolled repeated infections, or other serious uncontrolled concomitant diseases.
13. Moderate or severe renal damage [creatinine clearance ≤50ml/min (calculated according to Cockroft and Gault equation), or serum creatinine> ULN].
14. Acute or chronic active hepatitis B, hepatitis C infection, hepatitis B virus (HBV) DNA>2000IU/ml or 10^4 copies/ml, hepatitis C virus (HCV) RNA>10^3 copies/ml, hepatitis B surface antigen (HbsAg) is positive at the same time as anti-HCV antibody.
15. Allergic to any research drug ingredients.
16. Participating in other trials within 4 weeks before enrollment.
17. Not suitable to participate in this trial for any reason judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission rate | 4-month
  Completely resected tumor specimens and all sampled regional lymph nodes were detected without residual infiltration (ie ypT0 ypN0 in AJCC staging version 8.0)

SECONDARY OUTCOMES:
Objective response rate | 3-month
  Defined as the proportion of subjects whose best overall response is complete response (CR) and partial response (PR).
R0 resection rate | 4-month
  Defined as the proportion of patients who have achieved R0 resection. R0 surgery is defined as complete resection of the tumor without visible residual lesions either by naked eyes or under microscope.
3-year overall survival rate | 3-year
  Overall survival (OS) is defined as the time from the enrollment to death for any cause. The Kaplan-Meier curve of OS will be proformed to calculted the 3-year OS rate.
Progress-free survival | 3-year
  1) In patients who underwent radical surgery, the time from enrollment to recurrence or death; 2) in patients who did not undergo radical surgery, the time from enrollment to progression (according to RECIST 1.1) or death determined as disease progression.
3-year PFS rate | 3-year
  The Kaplan-Meier curve of progress-free survival will be proformed to calculted the 3-year PFS rate.

OTHER OUTCOMES:
Adverse events (AEs) | 4-month
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Li, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No